CLINICAL TRIAL: NCT03011983
Title: Neural Injury in Adolescents With Concussion
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: 16-013207
Record Dates: First submitted 2016-12-29; First posted 2017-01-06 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Mild Traumatic Brain Injury; Concussion, Mild; Acute Brain Injury
Keywords: Magnetoencephalography (MEG); Magnetic resonance imaging (MRI)
MeSH Terms: conditions — Brain Concussion; Brain Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Adolescents With Concussion: Adolescents with a concussion (n=120) will undergo neuroimaging (MEG and MRI) and neuropsychology assessments at two time points in the acute and chronic periods after injury, respectively. Brain imaging injury measures will be compared to a control normative database we will create. These brain measures will also be associated with cognitive and clinical outcomes.
  Interventions: Device: MEG; Device: MRI; Behavioral: Neuropsychology assessment
- Adolescents Without Concussion: Age- and gender-matched healthy controls (n=160) will be recruited to establish a normative database of whole-brain slow-wave maps from MEG resting-state data as well as white-matter diffusion measures from MRI.
  Interventions: Device: MEG; Device: MRI; Behavioral: Neuropsychology assessment

INTERVENTIONS:
Device: MEG — MEG is a non-invasive functional imaging technique that can measure slow-wave neural activity.
Device: MRI — MRI is a non-invasive imaging modality that provides measures of brain structure.
Behavioral: Neuropsychology assessment — A battery of tests will be administered by a neuropsychologist to evaluate the cognitive function of adolescents with concussion compared to healthy controls.

SUMMARY:
This study utilizes multimodal brain imaging to obtain quantitative biomarkers of brain injury and to improve understanding of the biological basis of brain pathology in adolescents with concussion. Adolescents with a concussion will undergo neuroimaging and neuropsychology assessments acutely and four months after injury.

DETAILED DESCRIPTION:
Concussion is a highly prevalent condition in adolescence, but it remains a clinical diagnosis that largely relies on subjective patient report with no reliable objective biomarkers for diagnosis. Traditional clinical brain imaging has not been found useful for concussion as the pathology is generally not visible on conventional acute MRI or CT. The proposed study addresses this gap in concussion diagnosis and management by examining the sensitivity of magnetoencephalography (MEG) for identifying areas of brain injury through detection of abnormal neural activity (slowing) in adolescents with concussion compared to healthy controls. Adolescents with a concussion will complete neuroimaging (MEG and MRI) and neuropsychology assessments at two time points within ten days and then again 4 months post-injury. Healthy controls will complete neuroimaging and neuropsychology assessments at a single time point.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of concussion and within 2 weeks of injury (case subjects)
* No history of diagnosed concussion (control subjects)

Exclusion Criteria:

* Head injury within 1 year of recent concussion (case subjects)
* History of neurologic, psychiatric, developmental or learning disorders (all subjects)

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Adolescents with a recent concussion will be recruited from outpatient clinics in orthopedics and trauma surgery. Healthy controls will be obtained via volunteers and previous brain imaging research studies.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Difference in MEG Whole-Brain Slow-Wave Sensitivity between Controls and Concussion Patients | Up to 2 months
  Whole-brain, resting-state slow-wave maps of whole brain activity will be obtained from the MEG imaging in both adolescents with a concussion and healthy controls. Control images will be analyzed to determine a whole brain z-score value that includes typically developing controls below the 95th percentile, the z-score threshold for this group). Z-score images for the adolescents with concussion will be obtained and the number of adolescents with concussion above this z-score threshold will be determined, and compared to the healthy controls. The sensitivity and specificity of this method determined.

SECONDARY OUTCOMES:
Difference in MRI White-Matter Diffusion Measures between Controls and Concussion Patients | Up to 2 months
  MRI diffusion data will be collected to examine associations between abnormal brain slowing and white matter damage in the adolescents with a concussion versus controls. Regions showing abnormal white matter diffusion will be comparing to normative control diffusion data.

CONTACTS AND LOCATIONS:
Overall Officials: Christina L Master, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang MX, Theilmann RJ, Robb A, Angeles A, Nichols S, Drake A, D'Andrea J, Levy M, Holland M, Song T, Ge S, Hwang E, Yoo K, Cui L, Baker DG, Trauner D, Coimbra R, Lee RR. Integrated imaging approach with MEG and DTI to detect mild traumatic brain injury in military and civilian patients. J Neurotrauma. 2009 Aug;26(8):1213-26. doi: 10.1089/neu.2008.0672. PMID 19385722
- [Background] Huang MX, Nichols S, Robb A, Angeles A, Drake A, Holland M, Asmussen S, D'Andrea J, Chun W, Levy M, Cui L, Song T, Baker DG, Hammer P, McLay R, Theilmann RJ, Coimbra R, Diwakar M, Boyd C, Neff J, Liu TT, Webb-Murphy J, Farinpour R, Cheung C, Harrington DL, Heister D, Lee RR. An automatic MEG low-frequency source imaging approach for detecting injuries in mild and moderate TBI patients with blast and non-blast causes. Neuroimage. 2012 Jul 16;61(4):1067-82. doi: 10.1016/j.neuroimage.2012.04.029. Epub 2012 Apr 20. PMID 22542638
- [Background] Lewine JD, Davis JT, Bigler ED, Thoma R, Hill D, Funke M, Sloan JH, Hall S, Orrison WW. Objective documentation of traumatic brain injury subsequent to mild head trauma: multimodal brain imaging with MEG, SPECT, and MRI. J Head Trauma Rehabil. 2007 May-Jun;22(3):141-55. doi: 10.1097/01.HTR.0000271115.29954.27. PMID 17510590
- [Background] Huang MX, Nichols S, Baker DG, Robb A, Angeles A, Yurgil KA, Drake A, Levy M, Song T, McLay R, Theilmann RJ, Diwakar M, Risbrough VB, Ji Z, Huang CW, Chang DG, Harrington DL, Muzzatti L, Canive JM, Christopher Edgar J, Chen YH, Lee RR. Single-subject-based whole-brain MEG slow-wave imaging approach for detecting abnormality in patients with mild traumatic brain injury. Neuroimage Clin. 2014 Jun 16;5:109-19. doi: 10.1016/j.nicl.2014.06.004. eCollection 2014. PMID 25009772